Comprehensive Home-based Self-management Support for COPD Patients PI: Dr. Alex D Federman

NCT04533412

Document Date: 9-06-2021

## STATISTICAL ANALYSIS PLAN

We compared the baseline characteristics of study participants in the intervention and control groups using a t-test, Wilcoxon Rank Sum test or chi-square test, as appropriate. We used a difference-in-differences (DiD) approach to examine the effects of intervention and control over time. Analyses were performed using generalized linear models with a REPEATED statement (SAS Proc GENMOD). As a feasibility trial, the study was not powered to detect statistically significant differences for outcomes between intervention and control arms, though P <0.05 was considered statistically significant for all outcomes analyses. All analyses were performed using SAS software, version 9.4 (SAS Institute, Inc., Cary, NC).